CLINICAL TRIAL: NCT05595135
Title: txt4AML: An Innovative Mobile Intervention to Improve Oral Anti-Cancer Medications Among Acute Myeloid Leukemia Patients
Brief Title: Mobile Intervention to Improve Adherence of Oral Anti-cancer Medications Among Acute Myeloid Leukemia Patients, the txt4AML Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: staffing
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 22D.340; JT 19501 (Other: JeffTrial Number)
Record Dates: First submitted 2022-10-18; First posted 2022-10-26 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Health services research (text messages, smart pill bottle) (Experimental): Patients receive interactive text messages to help with adherence to medications and a smart pill bottle with medication reminders on study.
  Interventions: Other: Text Message-Based Navigation Intervention; Other: Behavioral, Psychological or Informational Intervention; Other: Survey Administration; Other: Quality-of-Life Assessment

INTERVENTIONS:
Other: Text Message-Based Navigation Intervention — Receive interactive text messaging.
  Other Names: Automated Text Message-Based Navigation; Text Message-Based Navigation
Other: Behavioral, Psychological or Informational Intervention — Receive medication reminders via smart pill bottle
Other: Survey Administration — Ancillary studies
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment

SUMMARY:
This clinical trial studies how well a mobile intervention consisting of a text messaging program and an electronic "smart" pill bottle with medication reminders works to improve adherence to oral anti-cancer medications among patients with acute myeloid leukemia (AML). Medication adherence is how well patients take medications as prescribed by their doctors, and good medical adherence is when patients take medications correctly. Poor medication adherence has been shown to be a barrier to effective treatment. Collecting feedback on patient experiences using the mobile intervention may help doctors design new methods and material for providing educational information to AML patients who are taking oral anti-cancer medications.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To examine the feasibility, acceptability and preliminary efficacy of txt4AML in a pilot single arm study.

SECONDARY OBJECTIVE:

I. To explore the association between overall treatment responses and real-time oral anti-cancer medication (OAM) adherence.

EXPLORATORY OBJECTIVE:

I. To summarize and assess other patient-reported outcomes, collected either as patient chart review or through self-reported survey, as well as the patient post-intervention interviews.

OUTLINE:

Patients receive interactive text messages to help with adherence to medications and a smart pill bottle with medication reminders on study.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with acute myeloid leukemia (AML)
* Patients will be or is taking venetoclax (or any other oral anticancer medication) as part of their first line therapy
* Has a phone with text capabilities
* Among patients aged 18 and older we will enroll participants regardless of race or ethnicity

Exclusion Criteria:

* Individuals who are terminally ill (defined as having less than 2 months to live)
* Individuals for whom there is documentation of inability to provide consent in the medical record
* Do not speak/read English
* This study will exclude pediatric patients (defined as individuals under age 18 years)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-08-15 (Actual); Primary Completion 2023-05-05 (Actual); Study Completion 2023-05-05 (Actual)

PRIMARY OUTCOMES:
Real-time oral anticancer medication (OAM) medication adherence | At baseline
  Will be measured daily by AdhereTech wireless smart pill bottles, which are Health Insurance Portability and Accountability Act (HIPAA)-compliant Food and Drug Administration (FDA) Class I medical devices that monitor electronic tracking of bottle and percent of pills detected inside the bottle. Will be summarized using proportions and 95% Clopper-Pearson exact confidence intervals.
Real-time oral anticancer medication (OAM) medication adherence | at 1 month
  Will be measured daily by AdhereTech wireless smart pill bottles, which are Health Insurance Portability and Accountability Act (HIPAA)-compliant Food and Drug Administration (FDA) Class I medical devices that monitor electronic tracking of bottle and percent of pills detected inside the bottle. Will be summarized using proportions and 95% Clopper-Pearson exact confidence intervals.
Real-time oral anticancer medication (OAM) medication adherence | At 2 months
  Will be measured daily by AdhereTech wireless smart pill bottles, which are Health Insurance Portability and Accountability Act (HIPAA)-compliant Food and Drug Administration (FDA) Class I medical devices that monitor electronic tracking of bottle and percent of pills detected inside the bottle. Will be summarized using proportions and 95% Clopper-Pearson exact confidence intervals.
MD Anderson Symptom Inventory for acute myeloid leukemia/myelodysplastic syndrome (MDASI)-(AML)/MDS survey response | At baseline
  Will be analyzed using univariable logistic regression models with the primary predictor of averaged daily real-time OAM medication adherence.
MD Anderson Symptom Inventory for acute myeloid leukemia/myelodysplastic syndrome (MDASI)-(AML)/MDS survey response | At 1 month
  Will be analyzed using univariable logistic regression models with the primary predictor of averaged daily real-time OAM medication adherence.
MD Anderson Symptom Inventory for acute myeloid leukemia/myelodysplastic syndrome (MDASI)-(AML)/MDS survey response | At 2 months
  Will be analyzed using univariable logistic regression models with the primary predictor of averaged daily real-time OAM medication adherence.

SECONDARY OUTCOMES:
Complete remission (CR) | At baseline, 1, and 2 months
  Will be analyzed using univariable logistic regression models with the primary predictor of averaged daily real-time OAM medication adherence
Incomplete blood count recovery (Cri) | At baseline, 1, and 2 months
  Will be analyzed using univariable logistic regression models with the primary predictor of averaged daily real-time OAM medication adherence.
Partial remissions (PR) | At baseline, 1, and 2 months
  Will be analyzed using univariable logistic regression models with the primary predictor of averaged daily real-time OAM medication adherence.
Morphologic leukemia-free state (MLFS) | At baseline, 1, and 2 months
  Will be analyzed using univariable logistic regression models with the primary predictor of averaged daily real-time OAM medication adherence.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Sidney Kimmel Cancer Center at Thomas Jefferson University, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania